CLINICAL TRIAL: NCT01886014
Title: The Effect of Oxytocin on Placebo Analgesia: an Experimental Study in Healthy Volunteers Using a Double-blind Design
Brief Title: The Effect of Oxytocin on Placebo Analgesia: an Experimental Study in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Ulrike Bingel, PD Dr. Ulrike Bingel, attending of neurology, research group leader, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: placebo_oxy
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Mechanisms and Modulators of Placebo Analgesia in Healthy Volunteers
Keywords: pain; pain modulation; placebo analgesia
MeSH Terms: conditions — Pain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin (Experimental): application of intranasal oxytocin 40IE
  Interventions: Drug: Oxytocin
- placebo (Placebo Comparator): application of intranasal saline
  Both sprays (saline/oxytocin) are delivered in identical containers manufactured by the University pharmacy to assure blinding.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: oxytocin
Other: placebo
  Arms: placebo

SUMMARY:
Placebo responses contribute to medical treatment outcome. The purpose of this study is to determine whether a single intranasal application of oxytocin can increase the placebo response in an experimental model of placebo analgesia in healthy volunteers.

DETAILED DESCRIPTION:
Placebo responses contribute to medical treatment outcome. The purpose of this study is to determine whether a single intranasal application of oxytocin can increase the placebo response in an experimental model of placebo analgesia in healthy volunteers.

The rationale to study the effects of oxytocin on placebo analgesia is based on previous studies showing that oxytocin fosters processes such as empathy, trust and social learning, which are key elements of the patient-physician relationship that is pivotal to placebo responses. In this experimental mechanisms study we used oxytocin as a tool to modulate these factors.

Placebo analgesia is induced verbal instruction. Therefore two identically looking placebo ointments were applied to two sites of the participants' volar forearm. The ointments were introduced as a local anesthetic that could reduce or even abolish pain (placebo) and a control cream (control), respectively.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, male and female
* being German-speaking
* Agreeing to participate, verified by completion of informed consent

Exclusion Criteria:

* acute or chronic pain condition
* use of any concomitant medication except contraceptives
* currently pregnant (verified by urine pregnancy test) or lactating
* major mental disorder
* Inability to comply with the study procedures
* abnormal pain sensitivity as indicated by pain threshold
* alcohol intake within last 24 hours

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Placebo analgesic responses | ~ 45 min after appliction of oxytocin or saline
  In this study the placebo analgesic response is defined as the difference in pain rating (visual analogue scale [0-100]) to thermal painful stimulation on the forearm on the placebo site compared to a control site.

SECONDARY OUTCOMES:
pain rating on the control site | ~45 min after application
  VAS pain rating [0-100] in the control (non-placebo) condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Bingel, MD, PhD, Principal Investigator — Department of Neurology, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Neurology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Kessner S, Sprenger C, Wrobel N, Wiech K, Bingel U. Effect of oxytocin on placebo analgesia: a randomized study. JAMA. 2013 Oct 23;310(16):1733-5. doi: 10.1001/jama.2013.277446. No abstract available. PMID 24150470